CLINICAL TRIAL: NCT04991805
Title: Descriptive Study of the Incidence of Malignancy in Severe Asthma Patients Receiving Benralizumab and Other Biologic Therapy, a Post Authorization Safety Study
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D3250R00042; EUPAS26310 (Other: ENCePP)
Record Dates: First submitted 2021-07-28; First posted 2021-08-05 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Asthma; Neoplasms
MeSH Terms: conditions — Asthma; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (3):
- Benralizumab: Patients who have received Benralizumab.
- Other biologics: Patients who have received non benralizumab biologics.
- Non-biologic: Patients who have received non biologic drug.

SUMMARY:
This is a real-world, observational, prospective cohort study in patients with severe asthma recruited into the International Severe Asthma Registry (ISAR) and the US severe asthma registry (CHRONICLE) and followed-up for occurrence of new malignancies. The primary objective is to measure the incidence of malignancy in the overall severe asthma population as well as its relevant subgroups, including patients receiving benralizumab, patients receiving non-benralizumab biologics, and patients not receiving biologics. The secondary objective is to describe the clinical characteristics of new malignancy cases that develop in severe asthma patients and relevant subgroups.

ELIGIBILITY:
Inclusion Criteria:

* The study population includes patients with severe asthma recruited into ISAR and CHRONICLE. Severe asthma patients are defined as those receiving treatment consistent with Global Initiative for Asthma (GINA) Step 5 or who are uncontrolled on GINA Step 4 treatment regimens.

Exclusion Criteria:

- Patients who are not willing and able to sign written informed consent

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes patients with severe asthma recruited into ISAR and CHRONICLE. Severe asthma patients are defined as those receiving treatment consistent with Global Initiative for Asthma (GINA) Step 5 or who are uncontrolled on GINA Step 4 treatment regimens. The three main study groups are: severe asthma patients who receive benralizumab, who receive non-benralizumab biologics, and those who do not receive any biologics.
Sampling Method: Non-Probability Sample
Enrollment: 14000 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-04-05 (Actual)

PRIMARY OUTCOMES:
Neoplasm | Annually, up to 5 years
  Incidence of neoplasm each year, starting from index date.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian P.J. Rabe, DHPeD, MSc, MD, FRSPH, Principal Investigator — AstraZeneca
Locations (2):
- Research Site, Stockholm, Sweden
- Research Site, Norwich, Norfolk, United Kingdom

REFERENCES:
- See also: D3250R00042-pass-csp-v4_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3250R00042&attachmentIdentifier=1532d621-0985-4507-888c-fdf616382105&fileName=D3250R00042-pass-csp-v4_Redacted.pdf&versionIdentifier=
- See also: CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3250R00042&attachmentIdentifier=7108d299-a2a1-4aa0-a446-7f6c4b0070d4&fileName=Malignancy_PASS_CSR_Synopsis_(EUPAS26310_NCT04991805).pdf&versionIdentifier=